CLINICAL TRIAL: NCT06120972
Title: A Non-randomized Prospective Phase II Study of Upfront Maintenance Olaparib in Advanced Ovarian Cancer BRCAwt Patients With Known Homologous Recombination Deficiency
Brief Title: Upfront Maintenance Olaparib in Advanced Ovarian Cancer BRCAwt Patients With Known Homologous Recombination Deficiency
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated due to Olaparib losing patent
Sponsor: Alexander B Olawaiye, MD (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Alexander B Olawaiye, MD, Professor, Department of Obstetrics, Gynecology & Reproductive Sciences, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 22-066
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer
Keywords: BRCAwt; homologous recombination deficiency (HRD); PARP inhibitors; homologous recombination repair (HR)
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olaparib (maintenance) (Experimental): 300 mg Olaparib (tablets) will be taken orally, twice a day (approximately every twelve hours)
  Interventions: Drug: Olaparib tablet

INTERVENTIONS:
Drug: Olaparib tablet — Lynparza, is a medication for the maintenance treatment of BRCA-mutated advanced ovarian cancer in adults. It is a PARP inhibitor, inhibiting poly ADP ribose polymerase, an enzyme involved in DNA repair.
  Other Names: Lynparza

SUMMARY:
This is a prospective non-randomized efficacy trial of olaparib maintenance therapy after frontline treatment with platinum-based therapy in advanced ovarian cancer patients with BRCAwt, homologous recombination deficient (HRD) disease.

DETAILED DESCRIPTION:
The use of PARP inhibitors has revolutionized how we think of the BRCA mutated population of ovarian cancer patients. However, this population with BRCA mutation is not the only one with homologous recombination deficiencies (HRD). Examples of BRCAwt but HR deficient mutations (HRD) include: BRIP1, RAD51C/D, and CHEK2 as well as epigenetic changes like BRCA methylation. This study is designed to provide information on if BRCAwt, HRD patients with advanced ovarian cancer benefit from maintenance olaparib monotherapy after frontline treatment. PAOLA-1 showed that this population had improved PFS from the addition of olaparib to bevacizumab but there is currently no information on how this population does with olaparib alone. For this reason, a similar population to PAOLA-1 will be used in this study. This study is designed to fill an important gap in the data provided by PAOLA-1. It is now considered standard of care for patients with BRCAwt, HRD disease to receive maintenance PARPi either alone (e.g. niraparib) based of PRIMA or in combination with bevacizumab based of PAOLA-1. Therefore, there is little to no concern that patients will be missing out on potentially beneficial therapy that could impact their prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance score of 0, 1, or 2
2. Life expectancy ≥ 16 months
3. Normal organ and marrow function as defined below: - Absolute neutrophil count (ANC) ≥ 1.5 x 109 /L - Platelets ≥ 100 x 109 /L - Hemoglobin (Hgb) ≥ 8 g/dL (blood transfusions to reach this amount are allowed) Page 15 of 69 - Serum creatinine ≤ 1.5 mg/dL - Total serum bilirubin ≤ 1.5 x ULN -AST and ALT ≤ 2.5 x ULN
4. Histologically confirmed advanced BRCAwt+ ovarian cancer with known recombinant deficiency
5. Measurable disease per RECIST 1.1
6. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) or Clinical examination and, which is suitable for accurate repeated measurements. OR At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline using CT/MRI/plain x-ray and is suitable for repeated assessment.

Exclusion Criteria:

1. Previous enrollment in the present study
2. Participation in another clinical study with an investigational product (IP) in the last 3 months.
3. BRCA 1 or 2 germline mutation
4. Use of hyperthermic intraperitoneal chemotherapy as part of their upfront adjuvant therapy
5. Non-epithelial origin of the ovary, the fallopian tube or the peritoneum (ie germ cell tumors)
6. Ovarian tumors of low malignant potential (eg borderline tumors) or mucinous carcinoma
7. Synchronous primary endometrial cancer unless both of the following criteria are met:

   1. Stage <II
   2. Aged <60 years at the time of diagnosis of endometrial cancer with stage IA or IB grade I or II, or stage IA grade III endometrial carcinoma OR aged ≥60 years at the time of diagnosis of endometrial cancer with stage IA grade I or II endometrioid adenocarcinoma. Subjects with serous or clear cell adenocarcinoma or carcinosarcoma of the endometrium are not eligible
8. Other malignancy within the last 5 years except adequately treated non-melanoma skin cancer; curatively treated in situ cancer of the cervix; ductal carcinoma in situ. Subjects with a history of localized malignancy diagnosed over 5 years ago may be eligible provided they completed adjuvant systemic therapy prior to enrollment and remain free of recurrent or metastatic disease.
9. Subjects with a history of primary triple-negative breast cancer may be eligible provided they completed definitive anticancer treatment more than 3 years ago and remain breast cancer free prior to start of study treatment
10. Subjects with MDS/ AML history
11. Subjects who experienced, for at least one cycle, a delay of >2 weeks because of prolonged hematologic recovery during first-line chemotherapy
12. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment Major surgery within 4 weeks of starting study treatment; subjects must have recovered from any effects of any major surgery
13. Previous allogenic bone marrow transplantation or double umbilical cord blood transplantation (dUCBT).
14. Any previous treatment with poly(adenosine diphosphate-ribose) polymerase inhibitor, including olaparib
15. Administration of other simultaneous chemotherapy drugs, any other anticancer therapy or antineoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period (hormonal replacement therapy is permitted as are steroidal antiemetics)
16. Current or recent (within 10 days prior to enrollment) chronic use of aspirin >325 mg/day
17. Concomitant use of known strong cytochrome P450 3A4 (CYP3A4) inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib or study treatment is 2 weeks.
18. *Concomitant use of known strong (eg.e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg.e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib or study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
19. Clinically significant (eg active) cardiovascular disease, including:

    1. Myocardial infarction or unstable angina pectoris within ≤6 months of enrollment
    2. New York Heart Association grade ≥2 congestive heart failure
    3. Poorly controlled cardiac arrhythmia despite medication (subjects with rate controlled atrial fibrillation are eligible), or any clinically significant abnormal finding on resting electrocardiogram
    4. Peripheral vascular disease grade ≥3 (eg symptomatic and interfering with activities of daily living requiring repair or revision)
20. Previous cerebrovascular accident, transient ischemic attack or subarachnoid hemorrhage within 6 months prior to enrollment
21. History or evidence of hemorrhagic disorders within 6 months prior to enrollment
22. Evidence of bleeding diathesis or significant coagulopathy (in the absence of coagulation)
23. History or clinical suspicion of untreated brain metastases or spinal cord compression. Computed tomography (CT)/magnetic resonance imaging (MRI) of the brain is mandatory (within 4 weeks prior to enrollment) in the case of suspected brain metastases. Spinal MRI is mandatory (within 4 weeks prior to enrollment) in the case of suspected spinal cord compression
24. History or evidence upon neurological examination of central nervous system disease (eg uncontrolled seizures), unless adequately treated with standard medical therapy
25. Significant traumatic injury during 4 weeks prior to enrollment
26. Subjects with evidence of abdominal free air not explained by paracentesis or recent surgical procedure
27. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the subject at high risk for treatment related complications
28. Pregnant or lactating women
29. Subjects unable to swallow orally administered medication and subjects with gastrointestinal disorders likely to interfere with absorption of the study medication
30. Subjects with a known hypersensitivity to olaparib or any of the excipients of the product
31. Immunocompromised subjects, for example, with known active hepatitis (ie, hepatitis B or C) or subjects known to be serologically positive for human immunodeficiency virus.
32. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg.e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
33. Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
34. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
35. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no.7).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to progression (TTP) | Up to 12 months
  Time (median number of months) between enrolment and progression (defined by RECIST 1.1) or death, whichever occurs first, and censored at the last date of disease assessment in the absence of progressive disease. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
1-year Progression-free Survival (PFS) | Up to 12 months
  Percentage of participants free of disease progression at 1 year. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to 6 years
  Time (median number of months) between enrollment and progression or death, whichever occurs first, and censored at the last date of disease assessment in the absence of progressive disease. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Second Progression-free Survival (PFS2) | Up to 6 years
  Time (median number of months) between enrollment and second objective disease progression, or death from any cause, whichever occurs first, and censored at last date of disease assessment in the absence of second disease progression. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Overall Survival (OS) | Up to 6 years
  Time (median number of months) from enrolment to death from any cause and censored at date of last follow-up.
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC QLQ-C30) | At Baseline, Every 12 weeks during treatment, at End of Treatment, Up to 3 years
  The EORTC QLQ-C30 is a cancer-specific questionnaire assessing 15 health-related quality of life (HRQoL) scales through 30-items: a global health status, five functional scales (physical, role, emotional, cognitive, and social) and nine symptomatic scales (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). For each dimension, one score is generated on a 0-100 scale, with higher score representing better HRQoL. Minimal clinically important difference defined as ±10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander B Olawaiye, MD, Principal Investigator — UPMC Hillman Cancer Center

IPD SHARING:
Plan to Share IPD: No